CLINICAL TRIAL: NCT06325618
Title: Lymphedema, Low-grade Inflammation and the Vasculature in Turner Syndrome
Acronym: TSCOR_V
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-138-23
Record Dates: First submitted 2024-02-20; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-01

CONDITIONS: Turner Syndrome; Cardiovascular Diseases; Lymphedema; Inflammation
MeSH Terms: conditions — Turner Syndrome; Cardiovascular Diseases; Lymphedema; Inflammation | interventions — Indocyanine Green

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biopsies from skin, muscle, fat, urine, buccal swaps and blood will be analysed for DNA and RNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Turner Syndrome: Women with karyotype verified Turner Syndrome n=100
  Interventions: Other: No intervention other than obtaining biopsies; Drug: Indocyanine green (ICG)
- Female controls: Healthy, age-matched controls n=50
  Interventions: Other: No intervention other than obtaining biopsies; Drug: Indocyanine green (ICG)

INTERVENTIONS:
Other: No intervention other than obtaining biopsies — Skin, fat, and muscle biopsies will be obtained
Drug: Indocyanine green (ICG) — Indocyanine green will be injected to evaluate the lymphatic system.

SUMMARY:
100 women with karyotype verified TS, previously examined at 4 study visits during a 19-year period will be asked to participate in a 5th study visit. Healthy age-matched females will be included as controls in a ratio 2:1.

The aim is to examine and quantify the cardiovascular and lymphatic system in women with TS. The investigators will study a possible causal mechanism between the known pathologic phenotype and alterations in these systems to understand, prevent or treat the life-threatening complications in TS.

DETAILED DESCRIPTION:
Background:

Patients with Turner syndrome (TS) are at risk of many complications during childhood, adolescence, and adulthood, including reduced final height, estrogen deficiency, infertility, lymphedema, ischemic heart disease, aortic dilation and dissection, congenital heart defect, hypertension, stroke, and autoimmune diseases in general.

The aim of this study is to evaluate the lymphatic and cardiovascular system in a cohort of adult women with TS to elucidate any defects, abnormalities or dysfunctions that may explain the myriad of complications related to TS.

Hypotheses:

1. Both the lymphatic and cardiovascular system are affected in TS with alterations in both anatomy, flow, and function.
2. Changes in the lymphatic system are more prevalent than previously assumed, affecting both central and peripheral lymphatic vessels.
3. Changes in lymphatic transportation and development of cardiovascular malformations occur simultaneously in early fetal life, thus disease in either system may interplay with malfunctions in the other.
4. The vascular structure in both lymph- and cardiovascular tissue is affected throughout the body and low-grade inflammation could be a possible factor in this pathogenesis in TS.
5. Changes in the vascular structure affects flow through the systems resulting in increased stress point on vessel walls leading to a possible entry site for a dissection which can be detected through flow analyses.
6. Genomic examination of multiple tissues will help in understanding the underlying genomic background for the congenital malformations seen in TS

Design:

100 women with karyotype verified TS, previously examined at 4 study visits during a 19-year period will be asked to participate in a 5th study visit. Healthy age-matched females will be included as controls in a ratio 2:1.

The lymphatic system will be examined using three different techniques to assess changes in both anatomy and function.

1. The investigators will use Near infrared light to evaluate the lymphatic system and grade dysfunction and detect subclinical lymphedema. Indocyanine Green will be injected subcutaneously in the foot and hand and used to assess the flow 5-60 minutes after injection.
2. A novel MRI technique to illustrate slow moving fluids, thus visualizing lymphatic fluid, will be used to display the contrast between fluids and tissue to view the thoracic duct and more peripheral lymphatic vessels and quantify their function, abnormalities and morphology.
3. A DEXA scan will be performed to calculate and differentiate between subdermal fat and lymphatic drainage or edema.

To evaluate the cardiovascular system, the investigators will use MRI of the heart and aorta to asses both function and morphology to calculate, among others, mean cardiac output, stroke volume, ejection fraction and asses myocardial fibrosis. A novel technique is to use a PET-CT, as this has been associated with atherosclerosis, because it can visualize macrophage rich atherosclerotic plaques and thus detect otherwise undetectable low-grade inflammation and disease in the cardiovascular system which may contribute to the development of cardiovascular complications.

The investigators will also evaluate the flow in the aorta using 4D-flow measurements based on customized MRI protocols to evaluate stress on the aortic wall and analyze the risk of aortic wall rupture and dissection. The potential of this analysis is the possibility to identify patients at high risk and need for medical or surgical intervention at an early stage and thus prevent or minimize this acute life-threatening complication to TS.

Genomic studies: Samples will be taken from multiple tissues (Blood, fat, muscle, skin, buccal swaps, urine) and DNA and RNA will be isolated using standard methodology.

ELIGIBILITY:
Inclusion Criteria:

* Turner Syndrome

Exclusion Criteria:

* pregnancy
* contraindications for MRI

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Danish women.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Grade dysfunction of clinical and subclinical lymphedema using Indocyanine Green Lymphography and Magnetic Resonance Lymphangiography. | 3 year
  Lymphedema will be graded in a total score according to the International Society of Lymphology. The stages are: Stage 0: Subclinical lymphedema. • Stage 1: Early, reversible pitting edema. Stage 2: Irreversible lymphedema. Stage 3: End-stage lymphedema.
Detecting low-grade inflammation in Turner Syndrome preforming FDG-PET/CT-scans to locate low grade inflammation. | 3 years
Heat maps of the distribution of wall shear stress in the aorta | 3 years
  Using 4D-flow analyses heat maps of the aorta will be made to illustrate the distribution of wall shear stress.

SECONDARY OUTCOMES:
MRI evaluation and description of vascular abnormalities in Turner Syndrome | 3 years
  Aortic dimensions
Cardiac MRI to evaluate function | 3 years
  Diastolic and systolic function of the left ventricle
Cardiac MRI to evaluate fibrosis of the myocardium | 3 years
  Estimation of myocardial fibrosis
Mapping DNA-methylations patterns in multiple tissues | 3 years
  Mapping DNA-methylation patterns in muscle, skin, fat, blood and urine
Immunologic changes in Turner Syndrome | 3 years
  Measuring blood concentrations of neutrophiles and lymphocytes, to asses neutrophil-to-lymphocyte ratio (NLR).

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mortensen KH, Andersen NH, Gravholt CH. Cardiovascular phenotype in Turner syndrome--integrating cardiology, genetics, and endocrinology. Endocr Rev. 2012 Oct;33(5):677-714. doi: 10.1210/er.2011-1059. Epub 2012 Jun 15. PMID 22707402
- [Background] Hjerrild BE, Mortensen KH, Sorensen KE, Pedersen EM, Andersen NH, Lundorf E, Hansen KW, Horlyck A, Hager A, Christiansen JS, Gravholt CH. Thoracic aortopathy in Turner syndrome and the influence of bicuspid aortic valves and blood pressure: a CMR study. J Cardiovasc Magn Reson. 2010 Mar 11;12(1):12. doi: 10.1186/1532-429X-12-12. PMID 20222980
- [Background] Executive Committee. The Diagnosis and Treatment of Peripheral Lymphedema: 2016 Consensus Document of the International Society of Lymphology. Lymphology. 2016 Dec;49(4):170-84. PMID 29908550
- [Background] Yu DX, Ma XX, Zhang XM, Wang Q, Li CF. Morphological features and clinical feasibility of thoracic duct: detection with nonenhanced magnetic resonance imaging at 3.0 T. J Magn Reson Imaging. 2010 Jul;32(1):94-100. doi: 10.1002/jmri.22128. PMID 20578016
- [Background] Unno N, Nishiyama M, Suzuki M, Yamamoto N, Inuzuka K, Sagara D, Tanaka H, Konno H. Quantitative lymph imaging for assessment of lymph function using indocyanine green fluorescence lymphography. Eur J Vasc Endovasc Surg. 2008 Aug;36(2):230-236. doi: 10.1016/j.ejvs.2008.04.013. Epub 2008 Jun 4. PMID 18534875
- [Background] Mohanakumar S, Telinius N, Kelly B, Lauridsen H, Boedtkjer D, Pedersen M, de Leval M, Hjortdal V. Morphology and Function of the Lymphatic Vasculature in Patients With a Fontan Circulation. Circ Cardiovasc Imaging. 2019 Apr;12(4):e008074. doi: 10.1161/CIRCIMAGING.118.008074. PMID 30943769